CLINICAL TRIAL: NCT00890266
Title: Collagen Cross-linking With Riboflavin in a Hypotonic Solution, With UV Light, on Corneas Less Than 400 Microns Thick: an Exploratory Study.
Brief Title: Corneal Collagen Cross-linking With Hypotonic Riboflavin in Corneas Thinner Than 400 Microns
Acronym: HypotonicRibo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Peschke Meditrade, GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHAR1006; 08/H0721/15
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Keratoconus
Keywords: keratoconus; collagen cross-linking; riboflavin; UV light
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): Exploratory
  Interventions: Procedure: Collagen cross-linking with hypotonic riboflavin

INTERVENTIONS:
Procedure: Collagen cross-linking with hypotonic riboflavin — Topical anaesthesia, corneal epithelial debridement, application of hypotonic riboflavin 0.1% solution (20 minutes), application of UV light (30 minutes).
  Other Names: Medio-Cross® hypotonic solution

SUMMARY:
Corneal ectasia is a relative weakness in the structure of the cornea, which produces a progressive change in its shape which results in visual distortion. It is known that collagen cross-linking in the cornea occurs naturally with age, and in diabetes, both of which seem to prevent progressive ectasia. Corneal collagen cross-linking with riboflavin on corneas thicker than 400 microns has been shown to stabilize the cornea in keratoconus, and prevent progression of the disease.

The purpose of this study is to determine whether corneal collagen cross-linking with riboflavin in a hypotonic solution, with UV light, on corneas less than 400 microns thick, leads to stabilisation of corneal ectasia.

DETAILED DESCRIPTION:
When cross-linking corneas of > 400 microns, riboflavin in a solution with high molecular weight dextran T500 is used to prevent corneal swelling during the administration of the drops and the UV treatment. However if riboflavin is applied to a cornea in a hypotonic solution (saline), then transient corneal oedema is created with thickening of the corneal stroma. In this way it is thought that the temporarily thickened cornea can be treated with UV whilst still providing a sufficient thickness to absorb the UV to an extent that endothelial cell damage is avoided.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus
* Corneas thinner than 400 microns, but thicker than 250 microns

Exclusion Criteria:

* Evidence of other corneal disease in the eye to be treated (e.g., Herpes simplex keratitis)
* Women who are pregnant or nursing at the time of the initial treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04-22 (Actual); Primary Completion 2010-04-22 (Actual); Study Completion 2010-04-22 (Actual)

PRIMARY OUTCOMES:
Change in keratometry/corneal topography | 3 months

SECONDARY OUTCOMES:
Corneal endothelial cell count | 3 months
Visual acuity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chad K Rostron, FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Department at St George's Hospital, London, Greater London, United Kingdom

REFERENCES:
- [Background] Hafezi F, Mrochen M, Iseli HP, Seiler T. Collagen crosslinking with ultraviolet-A and hypoosmolar riboflavin solution in thin corneas. J Cataract Refract Surg. 2009 Apr;35(4):621-4. doi: 10.1016/j.jcrs.2008.10.060. PMID 19304080